CLINICAL TRIAL: NCT04861142
Title: Osteoporosis Treatment Protocol in Patients With Fragility Fractures: Application and Efficacy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University General Hospital of Heraklion (Other)
Responsible Party: Principal Investigator, Ioannis Daskalakis, Orthopaedic surgery resident, University General Hospital of Heraklion
Other Study IDs: 3224
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Patients adherent to the anti-osteoporotic medication
  Interventions: Drug: Anti-osteoporotic medication( alendronate or denosumab)
- Patients non-adherent to the anti-osteoporotic medication
  Interventions: Drug: Anti-osteoporotic medication( alendronate or denosumab)

INTERVENTIONS:
Drug: Anti-osteoporotic medication( alendronate or denosumab) — Initiation of anti-osteoporotic medication (alendronate or denosumab)

SUMMARY:
Osteoporosis and osteoporotic fractures, especially hip fractures, have a significant impact on public healthcare. Despite the fact that the patients that have suffered an osteoporotic fracture have 86% increased risk of sustaining a second osteoporotic fracture, the efforts to prevent these fractures remain inadequate. The in-hospital initiation of antiosteoporotic treatment in patients that have been admitted due to hip fracture has shown to improve treatment rates and contribute to second fracture prevention. For this purpose the Arbeitsgemeinschaft für Osteosynthesefragen (AO) Foundation has introduced an algorithm that can be used by Orthopedic surgeons for the prevention of second fracture in patients that have already suffered an osteoporotic fracture. The purpose of this thesis is to study the efficacy of this algorithm in preventing the second fracture in the greek population. The study will include patients that have been admitted in the Orthopedics department of the University Hospital of Heraklion due to hip fracture. Bone density measurement will be performed using the DXA method and antiosteoporotic treatment will be administered according to the algorithm. These patients will be included in the hip registry of the Orthopedics department and the follow-up will last for 2 years .The primary aims of the study are: a)evaluation of the adherence to the antiosteoporotic medication b)the efficacy of the adherence to the aforementioned clinical algorithm in the secondary fracture prevention in the greek population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hip fractures after low-energy falls(fragility fractures)

Exclusion Criteria:

-Patients with hip fractures after high energy falls

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hip fractures after low-energy falls (fragility fractures), that are operatively treated in our department.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Adherence to the prescribed anti-osteoporotic medication | 1 year
Secondary fracture incidence | 1 year

SECONDARY OUTCOMES:
Morbidity and mortality of operatively treated hip fractures in our department | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Daskalakis, Orthopaedic Surgery Resident, Principal Investigator — University Hospital of Heraklion; Theodoros Tosounidis, Assistant Professor, Study Director — University Hospital of Heraklion; Apostolos Karantanas, Professor, Study Chair — University Hospital of Heraklion; Georgios Kontakis, Professor, Study Chair — University Hospital of Heraklion
Locations (1):
- University Hospital of Heraklion, Heraklion, Crete, Greece